CLINICAL TRIAL: NCT03357640
Title: Are the Combined Oral Contraceptive Pills Needed for Management of the Simple Ovarian Cysts in Reproductive Women? (Randomized Controlled Study)
Brief Title: Are the Combined Oral Contraceptive Pills Needed for Management of the Simple Ovarian Cysts in Reproductive Women?
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid mohammed salama, assistent professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: khalid4
Record Dates: First submitted 2017-11-24; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Ovary Cyst
MeSH Terms: conditions — Ovarian Cysts

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Both trial participants and research coordinator will be blinded about the treatment after assignment. Oral contraceptive pills and placebo will be put in 2 packages with different colors and only the main researcher will know the type of treatment used for each group. Unbinding is only permissible, if sever morbidity or even mortality occur to any participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- no intervention (Placebo Comparator): The women will receive one package of placebo. They also will receive a diary card for recording oral contraception intake to be returned to the physician on the next period. An appointment for the women in this group will be scheduled at one month of treatment for the second ultra-sonography. If the ovarian cyst does not show remission, the women will continue the same treatment and will follow up in another month by transvaginal ultra-sound. If the ovarian cyst still persists or progresses at the second month, the women will be followed up for third month.
  Interventions: Drug: combined oral contraceptive pills
- combined oral contraception pills (Active Comparator): The women will receive intervention of one package of combined oral contraception pills and will be counseled about how to take oral contraception and informed of possible side effects. They also will receive a diary card for recording oral contraception intake to be returned to the physician on the next period. An appointment for the women in this group will be scheduled at one month of treatment for the second ultra-sonography. If the ovarian cyst does not show remission, the women will continue the same treatment and will follow up in another month by transvaginal ultra-sound. If the ovarian cyst still persists or progresses at the second month, the women will be followed up for third month.
  Interventions: Drug: combined oral contraceptive pills

INTERVENTIONS:
Drug: combined oral contraceptive pills — one package of oral contraception (Cilest containing norgestimate 250 microgram + ethinyl estradiol 35 microgram)
  Other Names: placebo

SUMMARY:
Women will be managed by either of the two modalities and will be followed up by transvaginal ultrasound monthly for three successive months to evaluate the size and location of the functional ovarian cyst (follicular), to compare the effect of different modalities of management whether remission, regression, progression or persistence of functional ovarian cyst.

The women will be assigned randomly to either study group to take oral contraceptive pills or to control group to take placebo. The 2 groups will be treated and followed up equally. Oral contraceptive pills will be given to the study group as follow:

The women will receive one package of oral contraception (Cilest containing norgestimate 250 microgram + ethinyl estradiol 35 microgram) and will be counseled about how to take oral contraception and informed of possible side effects. They also will receive a diary card for recording oral contraception intake to be returned to the physician on the next period. An appointment for the women in this group will be scheduled at one month of treatment for the second ultra-sonography. If the ovarian cyst does not show remission, the women will continue the same treatment and will follow up in another month by transvaginal ultra-sound. If the ovarian cyst still persists or progresses at the second month, the women will be followed up for third month. All results of the two groups will be compared. Data will be collected, tabulated according to the standard statistical method.

DETAILED DESCRIPTION:
Women will be managed by either of the two modalities and will be followed up by transvaginal ultrasound monthly for three successive months to evaluate the size and location of the functional ovarian cyst (follicular), to compare the effect of different modalities of management whether remission, regression, progression or persistence of functional ovarian cyst.

The women will be assigned randomly to either study group to take oral contraceptive pills or to control group to take placebo. The 2 groups will be treated and followed up equally. Oral contraceptive pills will be given to the study group as follow:

The women will receive one package of oral contraception (Cilest containing norgestimate 250 microgram + ethinyl estradiol 35 microgram) and will be counseled about how to take oral contraception and informed of possible side effects. They also will receive a diary card for recording oral contraception intake to be returned to the physician on the next period. An appointment for the women in this group will be scheduled at one month of treatment for the second ultra-sonography. If the ovarian cyst does not show remission, the women will continue the same treatment and will follow up in another month by transvaginal ultra-sound. If the ovarian cyst still persists or progresses at the second month, the women will be followed up for third month. All results of the two groups will be compared. Data will be collected, tabulated according to the standard statistical method.

ELIGIBILITY:
Inclusion Criteria:include women in reproductive age ovarian cysts unilateral, 2.5-6 centimeters in diameter, thin wall, unilocular without internal echoes and no solid parts.

-

Exclusion Criteria:

Exclusion criteria include premenarche, post menopause and neoplastic ovarian swelling (any swelling more than 6cm or multilocular).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 118 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Remission | 3 months
  The main outcome measure and was defined as ultrasonographic examination being unable to detect the ovarian cyst or the cyst being less than 2 centimeters in the largest dimension.

SECONDARY OUTCOMES:
Regression | 3 months
  Was defined as ultrasonographic examination being able to detect the same ovarian cyst at more than 2 centimeters in size, but with the largest dimension having decreased more than 50% of the pre-treatment measurement.
Progression | 3 months
  Was defined as ultrasonographic examination being able to detect the same ovarian cyst with the largest dimension having increased more than 25% of the pre-treatment measurement.
Persistence | 3 months
  Was defined as ultrasonographic examination being able to detect the same ovarian cyst with the same size or with a decrease in the largest dimension of less than 50% or an increase in the largest dimension of less than 25% of the pre-treatment measurement

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed K Alloush, Study Director — Benha University
Locations (1):
- Benha university, Banhā, Al Qalubia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided